CLINICAL TRIAL: NCT03711006
Title: The Effect of Fecal Microbiota Transplantation in Ulcerative Colitis - A Case Study
Brief Title: The Effect of Fecal Microbiota Transplantation in Ulcerative Colitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alice Højer Christensen (Other)
Responsible Party: Sponsor-Investigator, Alice Højer Christensen, Principal Investigator, MD, Ph.d., Senior Specialist in Medical Gastroenterology, Aleris-Hamlet Hospitaler København
Organization: Aleris-Hamlet Hospitaler København (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16049117
Record Dates: First submitted 2018-10-10; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Ulcerative Colitis
Keywords: Fecal Microbiota Transplantation
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: The trial is an open-label pilot study treating 7 patients with Ulcerative Colitis with 25 daily multi-donor FMT Capsules for 50 days with 6 months follow up including the treatment period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT treated patients (Experimental): Seven patients with active Ulcerative Colitis treated with 25 multi-donor FMT Capsules daily.
  Interventions: Other: Fecal Microbiota Transplantation Capsules

INTERVENTIONS:
Other: Fecal Microbiota Transplantation Capsules — 25 daily multi-donor FMT Capsules for 50 days
  Other Names: FMT Capsules

SUMMARY:
7 patients with active Ulcerative Colitis are treated with 25 multi-donor FMT Capsules daily for 50 days.

DETAILED DESCRIPTION:
7 patients with active Ulcerative Colitis are treated with 25 multi-donor FMT Capsules daily for 50 days All patients are followed with regular follow up after 2,4,8,12,16, 20 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Ulcerative Colitis (UC)
* SCCAI between 4 and 10 at inclusion
* On a stable dose of 5-aminosalicylic acid (5-ASA) or without current treatment.
* Previous treatment with glucocorticoids, thiopurines and/or biological treatment was accepted.
* Fecal Calprotectin > 250 mg/kg
* Colonoscopy performed within the last 3 years
* Capable of writing and speaking Danish
* Attending regular follow-ups by a specialist in gastroenterology.

Exclusion Criteria:

* Biological treatment within the last four weeks
* Treatment with antibiotics within 48 hours before intervention
* Alcohol use above current Danish guidelines (14 units/week for men and 7 units/week for women)
* Pregnancy or planned pregnancy
* Active cancer disease
* Medical treatment of mental disorder
* Other chronic gastroenterological disorder besides UC, Irritable Bowel Syndrome (IBS) or Reflux-disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Change in patient colitis symptoms as assessed using the Simple Colitis Clinical Activity Index (SCCAI) | Baseline, 2,8,16 and 24 weeks
  Simple Colitis Clinical Activity Index (SCCAI)

SECONDARY OUTCOMES:
Fecal microbiota biodiversity in patients with Ulcerative Colitis and difference to donors fecal microbiota diversity | Baseline
  Alpha diversity (Shannon-index)
Fecal microbiota biodiversity in fecal donors | At donor inclusion
  Alpha diversity (Shannon-index)
Changes in fecal microbiota biodiversity in patients with Ulcerative Colitis in comparison with value at baseline | 8, 16 and 24 weeks
  Alpha diversity (Shannon-index)
Changes in Fecal Calprotectin in the active treatment period and follow-up period | Baseline, 8,16 and 24 weeks
  Fecal Calprotectin
Changes in patient reported quality of life: IBDQ | Baseline, 8, 16 and 24 weeks
  Inflammatory Bowel Disease Questionnaire (IBDQ)

CONTACTS AND LOCATIONS:
Overall Officials: Alice H Christensen, MD, PhD, Principal Investigator — Aleris-Hamlet Hospitals Copenhagen
Locations (1):
- Aleris-Hamlet Hospital Copenhagen, Søborg, Denmark

IPD SHARING:
Plan to Share IPD: No
Data are available upon request